CLINICAL TRIAL: NCT04252729
Title: Effect of Psychotherapy on Quality of Life and Recurrence of Events in Patients With Recurrent Vasovagal Syncope: A Randomized Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauricio Ibrahim Scanavacca (Other)
Responsible Party: Sponsor-Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Clinical Unit Director, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4383/16/049
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Syncope
Keywords: Psychotherapy; Syncope; Quality of life; Psychoanalytic psychosomatics
MeSH Terms: conditions — Syncope | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychotherapy (Experimental): Psychotherapy sessions based on the theoretical line of Psychoanalytic Psychosomatics for 1 year, every 10 days.
  Interventions: Procedure: Psychotherapy
- No psychotherapy (No Intervention): Follow-up according to institutional routine, without psychotherapy sessions.

INTERVENTIONS:
Procedure: Psychotherapy — Psychotherapy sessions based on Psychoanalytic Psychosomatics
  Arms: Psychotherapy

SUMMARY:
Recurrent vasovagal syncope although presenting a benign prognosis in terms of survival, is associated with significant impairment of quality of life. The impaired emotional status is also related to the recurrence of the events, closing a negative cycle for the evolution of the disease. This study aims to evaluate the effect of psychotherapy on the quality of life and in the number of syncope and pre-syncope events during one year of follow-up of patients with recurrent vasovagal syncope.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vasovagal syncope with positive TILT TEST and recurrent episodes (≥2 episode within 6 months)
* Signed Free and Informed Consent Form

Exclusion Criteria:

* Severe comorbidity with life expectancy <1 year
* Age <18 years
* Current psychotherapeutic follow-up
* Cardiac or neurological syncope
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Quality of life analysis performed by the Short Form 36 Instrument | 1 week
  Data collected at first visit
Quality of life analysis performed by the Short Form 36 Instrument | 6 months
  Data collected at first visit, 6 and 12 months (global assessment and by specific domains).
Quality of life analysis performed by the Short Form 36 Instrument | 12 months
  Data collected at 12 months (global assessment and by specific domains).

SECONDARY OUTCOMES:
Demographic data | 12 months
  Gender, age, date of birth, race, monthly income and education level.
Number of comorbidities | 12 months
  Especially use of alcohol, drugs and smoking
Use of concomitant medication | 12 months
  Prescription medication that the participant uses.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Barros E Silva RLA, Volich RM, de Barros E Silva PGM, da Costa Darrieux FC, Scanavacca MI, Hachul DT. Effect of psychotherapy on recurrence of events and quality of life in patients with vasovagal syncope. Sci Rep. 2022 Apr 6;12(1):5745. doi: 10.1038/s41598-022-09513-1. PMID 35388029